CLINICAL TRIAL: NCT03623659
Title: Does Partial Zona Pellucida Removal From Vitrified-warmed Human Blastocysts Improve Delivery Rate in IVF? A Multicentric RCT on Laser Assisted Hatching
Brief Title: pArtiaL zonA pelluciDa Removal by assisteD hatchINg of Blastocysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Alessandra Alteri, Principal Investigator, PhD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALADDIN
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Infertility
Keywords: Assisted hatching; Zona pellucida; Implantation failure; Blastocyst; Cryopreservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AH group (Active Comparator): Subjects whose vitrified/warmed blastocysts will be subjected to the treatment of laser assisted hatching
  Interventions: Procedure: Laser assisted hatching
- Control group (No Intervention): Subjects whose vitrified/warmed blastocysts will be subjected to the same procedures except for the treatment of laser assisted hatching

INTERVENTIONS:
Procedure: Laser assisted hatching — After warming, blastocysts are subjected to laser assisted hatching (LAH) following the standard procedure.The LAH procedure lasts one minute per blastocyst.
  Arms: AH group

SUMMARY:
The aim of study is to assess the possible impact of assisted hatching on delivery rate after transfer of vitrified-warmed human blastocysts.

DETAILED DESCRIPTION:
Zona pellucida (ZP) manipulation, termed "assisted hatching" (AH), has been introduced in order to favor embryo hatching and ultimately improve assisted reproductive technology success but with poor proofs of safety and biological plausibility.

Vitrifying and warming of blastocysts may impair the successful hatching process of the embryo out of its ZP and its following implantation into the uterus. Theoretically, AH may facilitate the hatching process and subsequently increase implantation rates.

In this prospective randomized controlled trial (RCT), the hypothesis is to test whether the application of a partial AH to vitrified/warmed blastocysts might affect patients' delivery rate.

Patients with vitrified blastocysts will be randomized at the time of blastocyst warming to a study group (with AH) or a control group (without AH). AH will be performed at the expanded blastocyst stage using a laser technique and a laser opening will be initiated at the 1 o'clock position. Consecutive laser shots will be applied to reach the 5 o'clock position of the blastocyst. The blastocysts will then be cultured at least 2 h and subsequently transferred into the patient's uterus.

ELIGIBILITY:
Inclusion Criteria:

* single embryo transfer of vitrified/warmed blastocyst (SET)
* first or second frozen IVF (with or without Intracytoplasmic Sperm Injection) cycle of blastocysts
* first or second oocyte retrieval

Exclusion Criteria:

* Preimplantation Genetic Testing (PGT) cycle
* BMI > 35 kg/m2
* severe male factor
* abnormal uterine cavity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Delivery rate | 38 weeks after embryo transfer
  Number of deliveries, that result in a live birth, per transferred blastocyst

SECONDARY OUTCOMES:
Implantation rate | 6-7 weeks after transfer
  the number of gestational sacs observed at echographic screening at 6 weeks of pregnancy divided by the number of transferred embryos
Clinical Pregnancy rate | 4 weeks after transfer
  the ultrasonographic demonstration of an intrauterine gestational sac divided by the number of included women
Biochemical pregnancy rate | 4 week after transfer
  Pregnancies failing to progress to the point of ultrasound confirmation divided by the number of women with a positive pregnancy test on blood
Ongoing pregnancy rate | 20 weeks after transfer
  the ultrasonographic demonstration of an intrauterine gestational sac with fetal hearth divided by the number of included women
Multiple pregnancy rate | 4 week after transfer
  a pregnancy in which more than one fetus develops in the uterus at the same time divided by the number of women with a clinical pregnancy
obstetrical and neonatal complication rate | after birth; 9-10 months after transfer
  condition that adversely affects women and their foetal health during delivery
congenital anomalies rate | after birth, 9-10 months after transfer
  birth defects, congenital disorders, congenital malformations, or congenital abnormalities, are conditions of prenatal origin that are present at birth, potentially impacting an infant's health, development and/or survival divided by the number of livebirths

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Alteri, PhD, Principal Investigator — IRCCS San Raffaele
Locations (2):
- Italy (2):
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - IRCCS San Raffaele, Milan

REFERENCES:
- [Background] Alteri A, Vigano P, Maizar AA, Jovine L, Giacomini E, Rubino P. Revisiting embryo assisted hatching approaches: a systematic review of the current protocols. J Assist Reprod Genet. 2018 Mar;35(3):367-391. doi: 10.1007/s10815-018-1118-4. Epub 2018 Jan 19. PMID 29350315
- [Derived] Alteri A, Reschini M, Guarneri C, Bandini V, Bertapelle G, Pinna M, Rabellotti E, Ferrari S, Papaleo E, Paffoni A, Vigano P, Somigliana E. The effect of laser-assisted hatching on vitrified/warmed blastocysts: the ALADDIN randomized controlled trial. Fertil Steril. 2024 Jul;122(1):106-113. doi: 10.1016/j.fertnstert.2024.02.010. Epub 2024 Feb 9. PMID 38342371
- [Derived] Alteri A, Guarneri C, Corti L, Restelli L, Reschini M, Giardina P, Papaleo E, Somigliana E, Vigano P, Paffoni A. ALADDIN study: does assisted hatching of vitrified/warmed blastocysts improve live birth rate? Protocol for a multicentric randomised controlled trial. BMJ Open. 2020 Jul 19;10(7):e031544. doi: 10.1136/bmjopen-2019-031544. PMID 32690492